CLINICAL TRIAL: NCT05618470
Title: Randomized Controlled Clinical Study on Wumeiwan Jiawei Fang Use in Patients With Blepharospasm
Brief Title: Wumeiwan Jiawei Fang Use in Patients With Blepharospasm
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yang Wei, professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZZ11-040
Record Dates: First submitted 2022-10-21; First posted 2022-11-16 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Dry Eye Syndromes; Meige Syndrome; Blepharospasm; Hyperactivity
Keywords: Wumeiwan Jiawei Fang; Blepharospasm; Meige syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Meige Syndrome; Blepharospasm; Spasm | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wumeiwan Jiawei Fang (Experimental): This group will take Wumei pill granule orally.
  Interventions: Drug: Wumeiwan Jiawei Fang
- botulinum toxin A (Active Comparator): In this group, Botulinum toxin type A (Lanzhou Biopharmaceutical Co. LTD.) was injected locally around the eye.
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: Wumeiwan Jiawei Fang — orally administered Wumeiwan Jiawei Fang prescription granules, 1 dose a day, twice a day, once for 14 days, for 42 days.
  Other Names: nothing
  Arms: Wumeiwan Jiawei Fang
Drug: botulinum toxin A — Botulinum toxin (Lanzhou Biopharmaceutical Co., LTD.) was injected into the medial side of the upper eyelid, the lateral side of the upper eyelid, the lateral side of the lower eyelid, and the temporal orbicularis oculi muscle of the lateral canthus. The botulinum toxin type A was diluted into 50IU/ML with normal saline and injected with a 1ml skin test syringe (4\ 5-gauge needle), and 2.5IU was injected into each point. A total of 1 injection.
  Other Names: nothing
  Arms: botulinum toxin A

SUMMARY:
To evaluate the efficacy and safety of Jing Fang Wu Mei Wan Jiawei Fang in the treatment of idiopathic blepharospasm using a clinical randomized controlled trial method.

DETAILED DESCRIPTION:
Idiopathic blepharospasm is an idiopathic dysfunction characterized by involuntary spasms of the eyelids bilaterally that interfere with visual function and cause ocular discomfort. The incidence has increased each year in recent years, and the disease may present with persistent eye closure or even functional blindness in advanced stages. In some patients, the disease may be associated with submandibular dystonia, known as Meige's syndrome. Currently, the disease is treated symptomatically. Such as oral.These treatments not only have large side effects, but also make it difficult to relieve the patient of multiple lesions in the eyes, face and tongue. Chinese medicine has unique advantages in treating this disease, highlighting the overall diagnosis and solving different parts of the disease in an integrated manner. Wu Mei Wan is a traditional Chinese medicine prescription, and our team has been using Wu Mei Wan Jia Wei Fang for the treatment of Meige syndrome since 2009 under the leadership of Gao Jiansheng, a famous Chinese medicine teacher in the capital, and found significant therapeutic effects in preliminary clinical observation, but there is a lack of large sample of randomized controlled clinical studies. In this study, we propose to systematically observe the efficacy of traditional Chinese medicine in the treatment of idiopathic blepharospasm by using the traditional sutra formula for idiopathic blepharospasm as a test group and local botulinum toxin A injection as a control group, and to scientifically evaluate the efficacy of the Wu Mei Wan Jia Wei Fang in the treatment of idiopathic blepharospasm.The results were evaluated in order to provide new treatment options for the clinical management of idiopathic blepharospasm (including Meige syndrome) and to benefit more patients.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic blepharospasm met the diagnostic criteria.
2. The age ranges from 18 to 80 years.
3. Liver Yang deficiency,mixed syndrome of cold and heat.
4. Signed Informed consent

Exclusion Criteria:

1. Secondary blepharospasm due to keratoconjunctivitis, trichiasis, and blepharitis.
2. Open eyelid disuse.
3. hemifacial spasm.
4. The patient had undergone eye surgery in the previous 6 months.
5. Allergic to the ingredients in the medicine.
6. Corneal lenses were worn during the study.
7. A woman who is pregnant or breastfeeding.
8. Combined with cardiovascular, cerebrovascular,Liver and kidney function, hematopoietic system serious primary disease, mental patients, combined with stroke patients.
9. At the same time, use drugs that interfere with the evaluation of drug efficacy.
10. Idiopathic blepharospasm is treated with other drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-12 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The degree of relief of blepharospasm was evaluated by Jankovic Rating Scale. | Six months
  According to the Jankovic Rating Scale (JRS), in terms of severity and frequency, the score ranges from 0 to 4, with the highest score being 8. The higher the score is, the more severe the spasm is.
The Blepharospasm Disability Index (BSDI) was used to evaluate the impact of blepharospasm on daily living activities before and after treatment. | Six months
  A total of 6 items were included, including walking, reading, driving, shopping, watching television and general activities. Each item was scored from 0 to 4 points and was self-evaluated by the patients. The total score of BSDI was 24 points.The higher the score is, the more severe the spasm is.
Traditional Chinese Medicine（TCM） syndrome scale evaluated the change of systemic syndrome before and after treatment. | Six months
  The score for each syndrome is the sum of the highest scores obtained for each diagnosis of the syndrome. The full score is 30 points. Efficacy score = (Total score of pre-treatment symptoms➖Total post-treatment symptom score)/Total score of pre-treatment symptoms×100%. Symptoms basically disappear, reducing by 95 to 100 percent; Obvious effect: symptoms decreased significantly, reaching more than 75%; Effective: symptoms decreased to more than 55%; Ineffective: No or slightly reduced symptoms, only less than 50%..
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Six months
  According to whether there are common side effects of botulinum toxin such as ptosis, diplopia, photophobia, dry eye, gastrointestinal tract of exposed keratitis, whether there are gastrointestinal reactions and other side effects that may be related to the Chinese medicine granule preparation in this study.
According to the Jankovic rating scale, the recurrence was determined at 14 days, 42 days, 3 months and 6 months after medication | Six months
  According to the Jankovic rating scale, the recurrence situation at 14 days, 42 days, 3 months and 6 months after medication was determined, and the increase of spasm intensity by 1 grade or more was considered as recurrence.
Number of participants with treatment-related adverse events as assessed by systemic response, routine blood tests, liver function (ALT), kidney function (BUN, Cr). | Six months
  1. Systemic reaction (record at any time);
  2. Routine blood tests: the detection points were 14 days, 42 days, 3 months and 6 months after the first visit and treatment;
  3. Liver function (ALT), kidney function (BUN, Cr) : The detection points were 14 days, 42 days, three months and six months after the first visit and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: wei yang, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Eye Hospital, China Academy of Chinese Medical Sciences；GuangAnmen Hospital, China Academy of Chinese Medical Sciences；XiYuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China